CLINICAL TRIAL: NCT04666623
Title: IMPORTANCE Trial - A Provisional Study-design of a Single-center, Phase II, Double-blinded, Placebo-controlled, Randomized, 4-week Study to Compare the Efficacy and Safety of Intranasal Esketamine in Chronic Opioid Refractory Pain
Brief Title: Compare the Efficacy and Safety of Intranasal Esketamine in Chronic Opioid Refractory Pain
Acronym: IMPORTANCE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: investigator decision
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ch20Benitez2
Record Dates: First submitted 2020-12-02; First posted 2020-12-14 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Cancer Pain
Keywords: Esketamine; Pain measurement; Opioid refractory pain
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Intervention Model Description: placebo-controlled, double-blinded with two parallel groups, superiority trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All investigators, patients, care providers, outcome assessors, and study statisticians will remain blinded with respect to the treatment allocation. Allocation sequence will be concealed for everyone involved in the trial, except for the pharmacist and the nurse responsible for patient's allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intranasal esketamine (56mg) (Active Comparator)
  Interventions: Drug: esketamine nasal spray
- placebo (Placebo Comparator)
  Interventions: Drug: placebo nasal spray

INTERVENTIONS:
Drug: esketamine nasal spray — unlabeled nasal injectors, each device will deliver 28mg of esketamine in a 200 μL solution, so in order to achieve the 56mg dose two devices will be required. On each dosing day during the trial, participants will self-administer at 2 time points 1 spray of the nasal spray into each nostril. Each administration will be separated by 5 minutes. The participants will receive the intervention twice weekly for 4 consecutive weeks.
  Arms: intranasal esketamine (56mg)
Drug: placebo nasal spray — unlabeled nasal injectors, each device will deliver 28mg of placebo in a 200 μL solution, so in order to achieve the 56mg dose two devices will be required. On each dosing day during the trial, participants will self-administer at 2 time points 1 spray of the nasal spray into each nostril. Each administration will be separated by 5 minutes. The participants will receive the intervention twice weekly for 4 consecutive weeks.
  Arms: placebo

SUMMARY:
This study is to assess the efficacy and safety of a four-week treatment with intranasal esketamine (56 mg) twice a week combined with opioid analgesic and adjuvant standard therapy in the management of adult patients with severe and opioid refractory chronic cancer pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient with refractory cancer pain, this pain defined when:

  * Multiple evidence- based biomedical therapies used in a clinically appropriate and acceptable fashion have failed to reach treatment goals that mainly include adequate pain reduction and/or improvement in daily living functioning activities.
  * Patients' functional activities do not allow a quality of life which is acceptable and/or pharmaceutical therapies have resulted in intolerable adverse effects.
* Psychiatric disorders and psychosocial factors that could influence pain outcomes have been assessed and appropriately addressed
* Cancer pain classified as chronic (persistent or recurrent pain lasting longer than 3 months), and currently refractory despite optimized analgesic therapy including an opioid.

  • Optimized analgesic therapy is arbitrarily defined as: oral morphine equivalent of 60 mg/d or more (or another strong opioid at optimized dose) plus at least one adjuvant analgesic drug, for at least 2 weeks.
* No increase in baseline long acting opioid dose or addition of a new adjuvant analgesic drug within 2 weeks prior to study entry
* Ability to communicate the intensity of pain using the NPRS pain scale ranging from (0 as no pain to 10 with severe pain).
* Ability to give fully informed written consent.
* Expect survival more than 3 months.

Exclusion Criteria:

* History of allergy or intolerance to esketamine or ketamine.
* History of allergy to disinfecting products containing quaternary ammonium, who might be susceptible to be allergic to denatonium benzoate.
* Concomitant use of xanthine derivatives (e.g. aminophylline, theophylline), ergometrine, or monoamine oxidase inhibitors.
* Active nasal/sinus dysfunction (e.g. allergic or infectious rhinitis) or presence of any lesion of the nasal mucosa.
* Pregnancy, breastfeeding and women of childbearing potential not using a highly effective contraception method.
* Uncontrolled hypertension, arrhythmia, heart failure, or untreated coronary artery disease. History of transient ischemic attacks, stroke, neurovascular disease, hemorrhage, severe head injury, hydrocephalus or elevated intracranial pressure within the last 3 months.
* History of primary or metastatic malignant brain lesions (uncontrolled or without previous treatment).
* Known aneurysmal vascular disease (including thoracic and abdominal aorta, intracranial, and peripheral arterial vessels) or arteriovenous malformation
* Uncontrolled psychiatric illness with psychosis/ hallucination (e.g. schizophrenia, acute psychosis).
* Alcohol abuse, drug abuse/ dependence within the past 6 months as self-reported.
* Cirrhosis or severe hepatic impairment defined as 5-fold elevation of transaminases
* Uncontrolled hyperthyroidism.
* Globe injuries or increased intraocular pressure (e.g. glaucoma).
* History of ulcerative or interstitial cystitis.
* Subjects scheduled to receive radiotherapy (RT) to a site of pain during the study period, or who have received RT to a site of pain within 2 weeks before study entry.
* Subjects scheduled to undergo surgical treatment during the study period likely to affect pain.
* Subjects on or starting chemotherapy if there is a significant expectation of that therapy affecting pain.
* Subjects who have not provided signed informed consent form.
* Concomitant use of drugs moderately or severely affecting cytochrome P450 activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Change in the eleven point Numeric Pain Rating Scale (NPRS) | 4 consecutive weeks (from Baseline to week 4)
  Change in the eleven point Numeric Pain Rating Scale (NPRS): assess pain intensity at enrollment and at each visit. Patients will be asked to rate their weekly pain on a scale from 0 to 10 where 0 equals "no pain" and 10 equals "the worst pain they can imagine. NPRS will be taken for both, during physical activity and at rest.

SECONDARY OUTCOMES:
Rescue morphine use | 4 consecutive weeks (from Baseline to week 4)
  The use of morphine rescue (whether it will be reduced, no change, or increased). This will be monitored using either the Aircure artificial intelligence through a mobile application or personal diaries.
Change in Brief Pain Inventory (BPI) | 4 consecutive weeks (from Baseline to week 4)
  Patients' functional status and satisfaction will be measured by the change in Brief Pain Inventory (BPI). (0 = no pain; 10 = pain as bad as you can imagine); No scoring algorithm, but "worst pain" or the arithmetic mean of the four severity items can be used as measures of pain severity; the arithmetic mean of the seven interference items can be used as a measure of pain interference.
Change in Patient Health Questionnaire (PHQ9) | 4 consecutive weeks (from Baseline to week 4)
  Change in depression score using the Patient Health Questionnaire (PHQ9) at enrollment and at each visit. It scores each of the nine depression criteria as "0" (not at all) to "3" (nearly every day).
Change in Side Effect Rating Scale for Dissociative Anesthetics (SERSDA) | 4 consecutive weeks (from Baseline to week 4)
  Change in Side Effect Rating Scale for Dissociative Anesthetics (SERSDA) at enrollment and at each visit. It assesses fatigue, dizziness, headache, nausea, changes in vision and mood changes (0 = side effects absent and 4 = adverse effect is bothersome).

CONTACTS AND LOCATIONS:
Overall Officials: Benito Benitez, MD, Principal Investigator — University Hospital Basel, Klinik für Mund-, Kiefer- und Gesichtschirurgie
Locations (1):
- University Hospital Basel, Klinik für Mund-, Kiefer- und Gesichtschirurgie, Basel, Switzerland

REFERENCES:
- [Derived] Fernandes M, Schelotto M, Doldi PM, Milani G, Ariza Manzano AA, Perera Valdivia D, Winter Matos AM, Hamdy Abdelrahim Y, Hamad Bek SA, Benitez BK, Romanelli Tavares VL, Basendwah AM, Albuquerque Sousa LH, Xavier NF, Zertuche Maldonado T, Toyomi de Oliveira S, Chaker M, Menon Miyake M, Uygur Kucukseymen E, Waqar K, Alkhozondar OMJ, Bernardo da Silva R, Droppelmann G, Vaz de Macedo A, Nakamura R, Fregni F. IMPORTANCE trial: a provisional study-design of a single-center, phase II, double-blinded, placebo-controlled, randomized, 4-week study to compare the efficacy and safety of intranasal esketamine in chronic opioid refractory pain. F1000Res. 2021 Jan 22;10:42. doi: 10.12688/f1000research.27809.1. eCollection 2021. PMID 33732434